CLINICAL TRIAL: NCT05357638
Title: Physical Training for People With Parkinson's Disease and Multiple Sclerosis: Effect on Mind and Body
Acronym: HersenFIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Netherlands Brain Foundation (Other)
Responsible Party: Principal Investigator, Dr. Erwin E. H. van Wegen, Principal Investigator, Associate Professor Neurorehabilitation, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL78096.029.21
Record Dates: First submitted 2022-04-12; First posted 2022-05-03 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Parkinson Disease; Multiple Sclerosis
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Training Group 1 (n=16) (Experimental): High Intensity Interval Training
  Interventions: Behavioral: High Intensity Interval Training (HIIT)
- Physical Training Group 2 (n=16) (Experimental): Continuous Aerobic Training
  Interventions: Behavioral: Continuous Aerobic Training (CAT)
- Physical Training Group 3 (n=16) (Experimental): Movement Advice
  Interventions: Behavioral: Movement Advice

INTERVENTIONS:
Behavioral: High Intensity Interval Training (HIIT) — 8 weeks of HIIT, 2x/week for about 30 minutes/session on a cycle ergometer
  Arms: Physical Training Group 1 (n=16)
Behavioral: Continuous Aerobic Training (CAT) — 8 weeks of CAT, 2x/week for about 50 minutes/session on a cycle ergometer
  Arms: Physical Training Group 2 (n=16)
Behavioral: Movement Advice — Weekly step goal, monitored using an activity tracker, +3000 steps/day for 5 days/week, step goal is based on average step count in the 4 weeks of baseline prior to the intervention
  Arms: Physical Training Group 3 (n=16)

SUMMARY:
People with Parkinson's disease and Multiple Sclerosis experience disabling motor and non-motor symptoms, which respond insufficiently to medication. To adequately alleviate disease burden, physical training is increasing acknowledged as an assisting therapy; however, the optimal dose of exercise in unknown.

DETAILED DESCRIPTION:
Next to complex motor deficits, people with Parkinson's disease and Multiple Sclerosis experience highly disabling non-motor symptoms; for example, anxiety and depression, cognitive decline, fatigue, and sleep problems. Physical training is increasingly recognized as an assisting and, importantly, safe therapy for these patients to alleviate disease burden. However, the optimal dose (i.e., type, frequency, intensity, duration) of exercise has not yet been established. This study aims to investigate differences in response patterns of motor and non-motor symptoms, blood-based biomarkers of neuroplasticity and neurodegeneration, as well as functional brain connectivity to eight weeks of high intensity interval training [2x/week, ~30 min/session], continuous aerobic training [2x/week, ~50 min/session], or movement advice [+3000 steps/day for 5 days/week monitored with an activity tracker]. Frequently repeated assessment of outcomes measures will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease (PD) or Progressive Multiple Sclerosis (MS)
* Hoehn & Yahr stage <4 (PD), Expanded Disability Status Scale score <6 (MS)
* Anxiety and/or depressive symptoms; Hospital Anxiety and Depression Scale (HADS) score >=8 points on HADS-A and/or HADS-D
* Sufficient cognitive ability to understand training instructions; Montreal Cognitive Assessment score >21 points
* Able to participate in intensive physical training, no contra-indications for exercise
* Stable medication regime for at least 4 weeks prior to inclusion
* Age >=18 years

Exclusion Criteria:

* Participation in intensive exercise program in the month prior to inclusion
* Relapse in the month prior to inclusion (MS)
* Symptoms indicating cardiovascular, pulmonary, or metabolic disease or cardiovascular, pulmonary, or metabolic disease which are not under control with medication
* abnormal electrocardiography in rest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety and depressive symptoms | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on anxiety and depressive symptoms, measured by the Hospital Anxiety and Depression Scale

SECONDARY OUTCOMES:
Change in disease severity | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on disease severity, measured by the Unified Parkinson's Disease Rating Scale (Parkinson's disease) (total score range 0-199, higher score = worse) or Expanded Disability Status Scale (Multiple Sclerosis)
Change in cognitive function (i.e., ability to inhibit cognitive interference) | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on cognitive function, measured by the Stroop Color Word Test
Change in cognitive function (i.e., mental flexibility) | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on cognitive function, measured by the Trail Making Test
Change in cognitive function (i.e., range of cognitive operations: motor speed, attention, and visuoperceptual functions) | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on cognitive function, measured by the Symbol Digit Modalities Test
Change in fatigue | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on fatigue, measured by the Checklist Individual Strength fatigue sub-scale
Change in sleep quality | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on sleep quality, measured by the Insomnia Severity Index
Change in well-being | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on well-being, measured by the Parkinson's Disease Questionnaire (8 items) (Parkinson's disease) or Multiple Sclerosis Impact Scale (29 items) (Multiple Sclerosis)
Change in quality of life | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on quality of life, measured by the Short Form health survey (36 items)
Change in motor capacity (i.e., walking speed) | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on motor capacity, measured by the 10-Meter Walk Test
Change in motor capacity (i.e., lower extremity function, mobility, and fall risk) | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on motor capacity, measured by the Timed Up and Go test
Change in motor capacity (i.e., finger dexterity) | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on motor capacity, measured by the Nine Hole Peg Test
Change in activities of daily living | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on activities of daily living, measured by the Nottingham Extended Activities of daily living Index
Change in biomarkers of neuroplasticity in blood | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on biomarkers of neuroplasticity in blood, measured by Brain Derived Neurotrophic Factor concentration
Change in biomarkers of neurodegeneration in blood | Baseline (week 0), week 4, week 12, week 16
  The effect of physical training on biomarkers of neurodegeneration in blood, measured by Neurofilament Light concentration
Change in brain morphology | Week 4, week 12
  The effect of physical training on brain morphology, measured by structural magnetic resonance imaging (MRI)
Change in structural brain connectivity | Week 4, week 12
  The effect of physical training on structural brain connectivity, measured by diffusion MRI + free-water content
Change in brain connectivity | Week 4, week 12
  The effect of physical training on brain connectivity, measured by resting state functional MRI
Change in brain iron concentration in the Substantia Nigra | Week 4, week 12
  The effect of physical training on brain iron concentration in the Substantia Nigra, measured by Quantitative Susceptibility Mapping methodology
Change in brain neuromelanin content | Week 4, week 12
  The effect of physical training on brain neuromelanin content, measured by neuromelanin-sensitive MRI
Change in daily mood | Weekly assessment from baseline to week 16
  The effect of physical training on daily mood, measured by the Visual Analogue Scale (total sore range 0-10, higher score = better)
Change in daily anxiety | Weekly assessment from baseline to week 16
  The effect of physical training on daily anxiety, measured by the Visual Analogue Scale (total sore range 0-10, higher score = better)
Change in daily ability to concentrate | Weekly assessment from baseline to week 16
  The effect of physical training on daily ability to concentrate, measured by the Visual Analogue Scale (total sore range 0-10, higher score = better)
Change in daily fatigue | Weekly assessment from baseline to week 16
  The effect of physical training on daily fatigue, measured by the Visual Analogue Scale (total sore range 0-10, higher score = better)
Change in daily sleep quality | Weekly assessment from baseline to week 16
  The effect of physical training on daily sleep quality, measured by the Visual Analogue Scale (total sore range 0-10, higher score = better)

CONTACTS AND LOCATIONS:
Overall Officials: Erwin EH van Wegen, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VU medical center, Amsterdam, North Holland, Netherlands

REFERENCES:
- See also: Website of the trial — http://www.hersenfit.amsterdam